CLINICAL TRIAL: NCT00604123
Title: A Randomized, Double Blind, Placebo-Controlled, Parallel Group Study Evaluating Effects of Intranasal JNJ-17166864 on Symptoms of Allergic Rhinitis in Adult Men or Women Allergic to Mountain Cedar Pollen
Brief Title: A Study Evaluating Effects of Intranasal JNJ-17166864 on Symptoms of Allergic Rhinitis in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR014041; 17166864NAP2001 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2008-01-08; First posted 2008-01-30 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Allergic Rhinitis
Keywords: JNJ-17166864; allergic rhinitis; pharmacokinetics; biomarkers; rhinitis symptoms; mountain cedar pollen
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JNJ-17166864 (Experimental)
  Interventions: Drug: JNJ-17166864
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-17166864 — JNJ-17166864 0.5 mg per nostril twice daily for 2 weeks.
  Arms: JNJ-17166864
Drug: Placebo — Placebo nasal spray twice daily for 2 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the clinical effectiveness, safety and pharmacokinetics of JNJ-17166864 in patients with seasonal allergic rhinitis.

DETAILED DESCRIPTION:
The study is conducted to prove the hypothesis that JNJ-17466864, as compared to placebo, can provide a 16% or greater improvement in nasal symptoms of seasonal allergic rhinitis. This is a randomized, blinded, placebo-controlled, parallel-group, 2-center outpatient study in adult men or women who have seasonal allergic rhinitis and have 2 year history (or longer) of mild to moderate allergic reaction to mountain cedar pollen. The study will be conducted in mountain cedar pollen season. 72 qualified patients will be admitted to the single-blind 7-day Run-in Period (placebo twice daily) to establish the Baseline allergic rhinitis symptom scores. Patient eligibility to enter the double-blind treatment phase will be based on patients' baseline nasal symptom scores. At least 66 eligible patients whose daytime average nasal symptom scores (of nasal congestion, nasal itching, rhinorrhea, and sneezing) is 2 or greater, with the daytime nasal congestion symptom score 2 or greater, on at least 4 of the 7 Run-in days will be admitted to the double-blind treatment phase, and randomized to either the JNJ-17166864 or placebo treatment group. During the Treatment Phase, patients will self-administer study medication (0.5 mg JNJ-17166864 or placebo per nostril) twice daily for 2 weeks, record allergic rhinitis nasal and ocular symptom scores, and complete the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ), to establish the In-Treatment scores. Pharmacokinetic and biomarker samples will be collected during treatment phase. Throughout the study, safety and tolerability will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical history of seasonal allergic rhinitis with onset and offset of nasal allergy symptoms during each of the past 2 mountain cedar allergy seasons
* Have positive prick skin test reaction to mountain cedar allergen at screening or have a documented positive prick skin test within 12 months prior to entering the treatment phase
* Good general health on the basis of physical examination (including nasal examination), medical history, vital signs, and 12-lead ECG performed at screening and on Day -2
* Good general health on the basis of clinical laboratory tests performed at screening
* Have no history of recent (within 14 days prior to study drug administration on Day 1) common cold or recent (within 14 days prior to study drug administration on Day 1) occupational exposures to inhaled irritants (e.g., industrial gases, dusts, pesticides) with the exception of mountain cedar pollen
* Have no history of recurrent or frequent epistaxis or recent episodes (within 14 days prior to study drug administration on Day 1) of nose bleeding
* Non-smoker or non-tobacco user (not smoked cigarettes or used tobacco-containing or nicotine-containing products for at least 3 months prior to screening.

Exclusion Criteria:

* Have asthma (Note: subjects with mild intermittent asthma are allowed)
* Chronic or intermittent use of inhaled, oral, intramuscular, intravenous, and/or potent or super-potent topical corticosteroids
* Use of any antihistamines during the study
* Under immunotherapy with mountain cedar extract
* Using prohibited medications or not having adequate washout period (prior to the start of Run-in) as specified: Intranasal or systemic corticosteroids (1 month), Intranasal cromolyn (2 weeks), Intranasal or systemic decongestants (3 days), Intranasal or systemic antihistamines (7 days), Intranasal tryptans,e.g. sumatryptan nasal spray, Imitrex (3 days), Intranasal ergotamines, e.g. dihydroergotamine mesylate nasal spray, Migranol (7 days), Singulair (7 days), Niaspan® extended-release tablets, or immediate release niacin (10 days)
* Documented evidence of acute or significant chronic sinusitis, as determined by the individual investigator
* Chronic use of concomitant medications including prescription medications (e.g., tricyclic antidepressants) that would affect assessment of the effectiveness of the study medication within 14 days prior to study drug administration on Day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To determine the effect of twice daily dosing of intranasal JNJ-17166864, compared to placebo, on nasal symptoms of seasonal allergic rhinitis (nasal congestion, nasal itching, rhinorrhea, and sneezing) | allergic rhinitis symptom score during treatment phase (2 weeks)

SECONDARY OUTCOMES:
To assess safety, tolerability, and pharmacokinetics | pharmacokinetics and biomarker assessment during treatment phase (2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- San Antonio, Texas, United States